CLINICAL TRIAL: NCT05973721
Title: To Investigate the Clinical Efficacy and Safety of Phage Therapy for Chronic Constipation
Brief Title: Clinical Study of Phage Therapy for Chronic Constipation Efficacy and Safety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIB-phage
Record Dates: First submitted 2023-07-17; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Pib Specific Phage; Intractable Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phage treatment group (Experimental)
  Interventions: Biological: phage

INTERVENTIONS:
Biological: phage — The treatment group was given one phage each time, once a day for two weeks

SUMMARY:
The overall aim was to evaluate the efficacy of PiB-specific phages for the treatment of refractory constipation through clinical studies, primarily for the publication of scientific papers and to guide the development of phage therapies. The purpose of this study will be subdivided into three aspects from three aspects: target exposure level, target occupation, and functional effects after acting on the target, including:1) The distribution of PIB phage in the intestine of patients with refractory constipation;2) The killing effect of PIB phage on PIB bacteria in refractory constipation patients;And 3) therapeutic effect of PIB phage on patients with refractory constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18-70 years, with confirmed chronic constipation and positive fecal bacteria test for PIB, agreed to participate in this experiment and signed an informed consent.

Exclusion Criteria:

* Severe heart failure, hypertension, cerebrovascular disease (e.g. stroke, moyamoya disease, etc.); Secondary constipation caused by psychotropic drug abuse; Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
To observe the curative effect of PIB phage on refractory constipation by defecation behavior of patients. | Baseline and six months after treatment
  Defecation behavior: A questionnaire was designed according to Rome IV criteria, and the questionnaire was collected and recorded, including the number of spontaneous bowel movements per week, PAC-QoL score, PAC-SYM score and Bristol stool trait score
The concentration of phage in feces was detected to evaluate the survival and survival ratio of active phage in the intestinal tract of patients. | Baseline and 24-48 hours after phage administration (first bowel movement)
Real-time PCR was used to detect the nucleic acid of PIB bacteria and HPLC was used to detect the distribution of fecal PIB phage in the intestinal tract of patients with refractory constipation | Baseline and two weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Tian, Dr, Principal Investigator — Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China